CLINICAL TRIAL: NCT07389798
Title: Effect of Remimazolam TIVA-Flumazenil Anesthesia Guided by Different Target Bispectral Index in Short ENT Surgeries: A Retrospective Cohort Study
Brief Title: Remimazolam TIVA-Flumazenil Anesthesia in Short ENT Surgeries
Acronym: TIVA
Status: Not yet recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, aijun xu, Professor, Tongji Hospital
Other Study IDs: RTFA
Record Dates: First submitted 2026-01-21; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Remimazolam; Total Intravenous Anesthesia; Bispectral Index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- AB group: Intraoperative BIS values ≤60
- HB group: Intraoperative BIS values >60

SUMMARY:
This study plans to categorize patients who underwent short-duration ENT surgeries with remimazolam TIVA combined with flumazenil antagonism based on whether their intraoperative BIS values were maintained below 60.

DETAILED DESCRIPTION:
This study plans to categorize patients who underwent short-duration ENT surgeries with remimazolam TIVA combined with flumazenil antagonism into two groups based on whether their intraoperative BIS values were maintained below 60. It aims to compare the differences in postoperative recovery quality between the groups, thereby providing evidence-based support for determining the optimal BIS target range during remimazolam TIVA.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* ASA I-III
* Underwent short-duration ENT surgery
* Underwent remimazolam TIVA combined with flumazenil antagonism.
* Continuous intraoperative BIS monitoring

Exclusion Criteria:

* Comorbid severe underlying diseases
* Intraoperative BIS data were missing or incompletely recorded
* Severe lack of medical records

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent short-duration surgeries with remimazolam TIVA combined with flumazenil antagonism in the Department of Otorhinolaryngology at Tongji Hospital, affiliated with Tongji Medical College, Huazhong University of Science and Technology, from January 1, 2024, to December 31, 2025, were included.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of intraoperative awareness | 2hours
  Modified Brice Interview From the start of surgery to the end of surgery

SECONDARY OUTCOMES:
Incidence of secondary sedation | 1 day
  Incidence of secondary sedation from flumazenil antagonization to discharge from the PACU
mean arterial pressure | 2 hours
  The fluctuation range of intraoperative mean arterial pressure during surgery
heart rate | 2 hours
  The fluctuation range of intraoperative heart rate during surgery
usage of vasoactive drugs | 2 hours
  Intraoperative use of vasoactive drugs during surgery
Drug doses | 2 hours
  Drug doses during surgery
Awakening time | 1 hours
  From the end of anesthesia to awakening.
PACU stay | 1 hours
  From admission to the PACU to discharge from the PACU.

CONTACTS AND LOCATIONS:
Overall Officials: Aihua Du, Dr, Study Chair — Tongji Hospital

IPD SHARING:
Plan to Share IPD: No
individual participant data (IPD) available to other researchers could be gotten from the PI Dr. aijun XU